CLINICAL TRIAL: NCT00876408
Title: Review of Molecular Profiling-Real Time Polymerase Chain Reaction (Rt-Pcr) in Unknown Primary Cancer: Role in Clinical Management and Primary Site Prediction
Brief Title: Review of Molecular Profiling-Real Time Polymerase Chain Reaction (Rt-Pcr) in Unknown Primary Cancer
Status: Completed | Type: Observational
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Biotheranostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SCRI OUTCOMES 08
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Unknown Primary Cancer
Keywords: RT-PCR molecular profiling assay; Molecular Profiling-Real Time Polymerase Chain Reaction; Unknown Primary; UPC; CUP
MeSH Terms: conditions — Neoplasms, Unknown Primary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This will be a retrospective review of 30 patients with unknown primary cancer who have had commercially available RT-PCR assays performed on biopsied tumors, in order to determine if the assay results are consistent with clinical features and useful for planning initial therapy or changing therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RT-PCR testing completed since commercialization of the RT-PCR assay in 2007.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 30 patients at Tennessee Oncology with unknown primary cancer have had commercially available RT-PCR assays done on their tissue biopsy since the assay became available in 2007. These patients are the subjects of this review.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To correlate the tissue of origin predicted by the RT-PCR assay with clinical and pathologic features of patients with carcinoma of unknown primary site. | 6 months

SECONDARY OUTCOMES:
To correlate the tissue of origin predicted by the RT-PCR with actual primary sites found subsequently in a subset of patients. | 6 months
To evaluate the utility of RT-PCR assay results in guiding treatment selection in patients with carcinoma of unknown primary site. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Greco, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States